CLINICAL TRIAL: NCT01245595
Title: A Randomized Placebo Controlled Trial of Aminophylline to Prevent Acute Kidney Injury in Children After Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: Aminophylline to Prevent Acute Kidney Injury in Children After Cardiac Surgery
Acronym: KIDPROAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, David Axelrod, MD, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18977
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury (AKI); Cardiopulmonary bypass (CPB)
MeSH Terms: conditions — Acute Kidney Injury | interventions — Aminophylline; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aminophylline (Active Comparator): Patients to receive aminophylline 5 mg/kg IV bolus then 1.8 mg/kg IV Q6 hours
  Interventions: Drug: Aminophylline
- Placebo (Placebo Comparator): Normal Saline Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aminophylline — 5 mg/kg IV bolus then 1.8 mg/kg IV Q6 hours
  Other Names: treatment
  Arms: Aminophylline
Drug: Placebo — Normal Saline
  Arms: Placebo

SUMMARY:
Children with congenital heart defects often need cardiac surgery with cardiopulmonary bypass (the "heart-lung machine"). Approximately 35 to 50% of these children will have "acute kidney injury," or damage to the kidneys, after the procedure. We currently have few medications to prevent this kidney injury. The hypothesis of this study is that giving aminophylline after heart surgery can decrease the acute kidney injury.

DETAILED DESCRIPTION:
Patients are randomized to receive aminophylline or placebo for 72 hours, in a blinded fashion. Serum theophylline levels monitor for safety of aminophylline dose. Goal theophylline levels is 5-7 mcg/ml. Laboratory results will be faxed directly to the pharmacy who will adjust subsequent aminophylline dosing to maintain appropriate theophylline levels. Urine output and serum creatinine levels will be monitored to assess acute kidney injury. Serum Neutrophil Gelatinase Associated Lipocalin (NGAL) levels will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Less than 18 years old, undergoing cardiac surgery with bypass
* neonates must be at least 36 weeks gestational age

Exclusion Criteria:

* History of arrythmia or seizure, on extracorporeal membrane oxygenation (ECMO) support, already taking aminophylline/theophylline, liver failure, sepsis, on renal replacement therapy

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2010-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: david m axelrod, md, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Childrens' Hospital, Palo Alto, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aminophylline | Placebo
Started | 72 | 72
Completed Full Course of Study Drug | 57 | 61
Completed | 72 | 72
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aminophylline | Placebo | Total
Number analyzed (Participants) | 72 | 72 | 144
Age, Continuous [Median (Inter-Quartile Range); unit: days] — Age, continuous, Days
  days | 154 [64 to 656] | 165 [58 to 1332] | 155 [60 to 1039]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 30 | 63
  Male | 39 | 42 | 81
Region of Enrollment [Number; unit: participants]
  United States | 72 | 72 | 144

OUTCOME MEASURES:

1. Primary Outcome: Acute Kidney Injury Measured by Kidney Diseases: Improving Global Outcomes (KDIGO) AKI Serum Creatinine Criteria
Description: Acute Kidney Injury measured by Kidney Diseases: Improving Global Outcomes (KDIGO) AKI Serum Creatinine criteria; KDIGO Stage is a measure of acute kidney injury.
Time Frame: 5 days
Measure: Number; unit: participants
Groups:
- Aminophylline: Patients to receive aminophylline 5 mg/kg intravenous (IV) bolus then 1.8 mg/kg IV every six (Q6) hours
  Aminophylline: 5 mg/kg IV bolus then 1.8 mg/kg IV Q6 hours
Arm/Group | Aminophylline | Placebo
Number analyzed (Participants) | 72 | 72
participants | 43 | 36

ADVERSE EVENTS:
Time Frame: Data were collected over the first five postoperative hospital days.
Description: Systematic Assessment: each patient was evaluated daily for an adverse event.
Arm/Group | Aminophylline | Placebo
Serious Adverse Events (participants affected / at risk) | 1/72 | 2/72
Other Adverse Events (participants affected / at risk) | 10/72 | 11/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aminophylline (N=72) | Placebo (N=72)
Low Cardiac Output requiring Cardiopulmonary resuscitation or Extracorporeal Membrane Oxygenation (Cardiac disorders) | 1 | 1
Cardiac Arrhythmia Leading to Cardiopulmonary Resuscitation (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aminophylline (N=72) | Placebo (N=72)
Accelerated Junctional Rhythm (Cardiac disorders) | 2 | 0
Junctional Ectopic Tachycardia (Cardiac disorders) | 4 | 2
Ventricular Tachycardia (Cardiac disorders) | 1 | 0
Ectopic Atrial Tachycardia (Cardiac disorders) | 0 | 2
Sinus Tachycardia (Cardiac disorders) | 1 | 1
Unspecified Tachycardia (Cardiac disorders) | 1 | 1
Acute Kidney Injury (AKI) (Renal and urinary disorders) | 1 | 1 — Managing physician treated AKI with aminophylline out of protocol
Pulmonary Hypertension with low cardiac output (Cardiac disorders) | 0 | 1
Bleeding (Blood and lymphatic system disorders) | 0 | 1
sepsis (Infections and infestations) | 0 | 1
Arm and jaw pain (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No